CLINICAL TRIAL: NCT04521907
Title: Correlative Study on Incidence and Risk Factors of Glaucoma-related Adverse Event at Various Durations After Congenital Cataract Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Other Study IDs: GRAE2 -zzh
Record Dates: First submitted 2020-08-12; First posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: The Incidence and Risk Factors of Glaucoma After Congenital Cataract Surgery
Keywords: Glaucoma; Incidence; Congenital cataract surgery
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Group 1 includes patients who underwent cataract surgery with primary IOL implantation
- Group 2: Group 2 includes patients who underwent cataract surgery with secondly IOL implantation
- Group 3: Group 3 includes patients who underwent cataract surgery without IOL implantation.

SUMMARY:
A retrospective chart review of 264 eyes from 177 patients was performed who underwent congenital cataract surgery before the age of 14 years. All patients' surgery was performed by the same experienced surgeon at the Eye Hospital of Wenzhou Medical University from May 2011 to March 2019. We recorded patient demographics and incidence and risk factors for glaucoma-related adverse event. This study to identify the incidence of and risk factors associated with postoperative glaucoma at various durations after congenital cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent lensectomy combined with limited anterior vitrectomy, with or without IOL implantation for congenital cataract, all by one surgeon

Exclusion Criteria:

* Patient had a preoperative IOP above 21mmHg, glaucoma, coexistent uveitis, metabolic syndromes/diseases or exposure to radiation.

Ages: 1 Month to 14 Years | Sex: All
Age Groups: Child
Study Population: Patients who underwent congenital cataract surgery at Eye hospital of Wenzhou Medical University
Sampling Method: Probability Sample
Enrollment: 177 (Estimated)
Dates: Start 2011-05-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of glaucoma after congenital cataract surgery | 2020.6.30
  The incidence of glaucoma at various durations after congenital cataract surgery
Demographic data, including sex, age at surgery, gestational history, family history of cataract, and laterality of disease, were collected. | 2020.6.30
  Risk factors

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmology and Optometry Hospital, Wenzhou, Zhejiang, China